CLINICAL TRIAL: NCT02893696
Title: The Effect of Sitting After Spinal Injection of Hyperbaric Local Anesthetic on Fetal Acid-base Balance After Cesarean Delivery
Brief Title: Extra Sitting Time After Spinal Anesthesia for Cesarean Section and Fetal Well-being
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no enrollment
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU012016-059
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Complications; Cesarean Section; Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediately Supine Position (Active Comparator): Women placed in supine position within 30 seconds after spinal injection of local anesthetic drug.
  Interventions: Other: Various sitting time
- Delayed Supine Position (Active Comparator): Women placed in supine position after three minutes of seating after spinal injection of local anesthetic drug.
  Interventions: Other: Various sitting time

INTERVENTIONS:
Other: Various sitting time — Various sitting time

SUMMARY:
After injection of the spinal anesthetic drug, women will be allowed to lie down immediately (0-30 sec) or after three minutes (180 sec) of sitting. The incidence of maternal hypotension and fetal umbilical cord blood pH will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Women with elective cesarean delivery at 39-42 wks gestation.

Exclusion Criteria:

* Women who shorter than 5'0" in height, those with primary or pregnancy-induced hypertension, macrosomia, multiple gestation will be excluded.
* Women with known risks of bleeding or potential hysterectomy such as those with placenta previa or accrete will also be excluded.
* If the epidural catheter cannot be placed within the specific time frame after the spinal injection, the case will be excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of fetal umbilical artery pH below 7.20 | At fetal delivery

SECONDARY OUTCOMES:
Incidence of maternal hypotension | During cesarean surgery

CONTACTS AND LOCATIONS:
Overall Officials: Weike Tao, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No